CLINICAL TRIAL: NCT02494739
Title: Investigation of the Antioxidant and Anti-inflammatory Effects of Yogurt Enriched With Polyphenols
Brief Title: Antioxidant and Anti-inflammatory Effects of Yogurt Enriched With Polyphenols
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Athanasios Z. Jamurtas, Associate Professor, University of Thessaly
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: UniYog-2015x
Record Dates: First submitted 2015-06-25; First posted 2015-07-10 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Oxidative Stress; Inflammation
Keywords: antioxidant; oxidative stress; inflammation; polyphenols; yogurt
MeSH Terms: conditions — Inflammation | interventions — Polyphenols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yogurt enriched with polyphenols (Experimental): Two yogurts (400g) enriched with polyphenols (10mg/100g yogurt) per day, for two weeks.
  Interventions: Other: Yogurt enriched with polyphenols
- Yogurt not enriched with polyphenols (Placebo Comparator): Two yogurts (400g) not enriched with polyphenols per day, for two weeks.
  Interventions: Other: Yogurt not enriched with polyphenols

INTERVENTIONS:
Other: Yogurt enriched with polyphenols — Yogurt enriched with polyphenols extracted from grape seeds
  Arms: Yogurt enriched with polyphenols
Other: Yogurt not enriched with polyphenols — Yogurt not enriched with polyphenols
  Arms: Yogurt not enriched with polyphenols

SUMMARY:
The purpose of this study is to investigate the possible antioxidant and anti-inflammatory effects of yogurt enriched with polyphenols after 2-week consumption by healthy individuals.

DETAILED DESCRIPTION:
Eighteen healthy adult volunteers of both sexes consumed yogurt (400g per day) enriched with polyphenols (10mg/100g yogurt) or yogurt (400g per day) not enriched with polyphenols for two weeks in a double-blind, crossover, randomized manner.There was a washout period of at least 10 days. Physiological data and blood samples were collected before and after consumption of each yogurt.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals
* Non-smokers

Exclusion Criteria:

* Current use of dietary supplements or drugs
* Metabolic disease
* Lactose intolerance
* Pregnant, pregnancy intention or breast feeding

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2015-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Antioxidant effects | Two weeks
  Indices of blood antioxidant status
Anti-inflammatory effects | Two weeks
  Indices of inflammation in blood

SECONDARY OUTCOMES:
Body composition | Two weeks
  Body fat percentage
Blood pressure | Two weeks
  Blood pressure at rest
Hydration | Two weeks
  Urine specific gravity
Resting heart rate | Two weeks
  Resting heart rate
Blood glucose levels | Two weeks
Triglyceride levels | Two weeks
Total cholesterol levels | Two weeks
High Density Lipoprotein cholesterol levels | Two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Athanasios Z Jamurtas, PhD, Study Director — University of Thessaly
Locations (1):
- Department of Physical Education & Sport Science of the University of Thessaly, Trikala, Karyes, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Najgebauer-Lejko D, Grega T, Tabaszewska M. Yoghurts with addition of selected vegetables: acidity, antioxidant properties and sensory quality. Acta Sci Pol Technol Aliment. 2014 Jan-Mar;13(1):35-42. doi: 10.17306/j.afs.2014.1.3. PMID 24583382
- [Background] Lamothe S, Azimy N, Bazinet L, Couillard C, Britten M. Interaction of green tea polyphenols with dairy matrices in a simulated gastrointestinal environment. Food Funct. 2014 Oct;5(10):2621-31. doi: 10.1039/c4fo00203b. Epub 2014 Aug 26. PMID 25154916